CLINICAL TRIAL: NCT01827995
Title: Simplified Medical Abortion in Rural India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristina Gemzell Danielsson, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WDuo2013
Record Dates: First submitted 2013-04-03; First posted 2013-04-10 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Pregnancy
Keywords: Low sensitivity urinary hCG; follow up; medical abortion; rural India; RCT
MeSH Terms: interventions — Diagnostic Self Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duo test (Other): Self assessment
  Interventions: Other: Self assessment
- Routine follow up (Other): Follow up in the clinic
  Interventions: Other: Routine assessment

INTERVENTIONS:
Other: Self assessment — Intervention group: Simplified followup Mifepristone at outpatient clinic, followed by the administration of misoprostol 24-48 hours later (in the clinic or at home). The women will not return to the clinic for routine follow up visit, but are given instructions on how to use a checklist and a low sensitivity pregnancy test around day 10-14. They are asked only to return if they have any health problems or screen positively. The low sensitivity urinary-hCG (with HCG of 1000 IU/ml) test will be used. Women will be provided the pregnancy test free of cost along with a pictorial checklist. A research assistant or a nurse will explain in detail how to use the pregnancy test as well as the checklist, and provide phone numbers in case of any questions or doubts. Follow-up interviews will be conducted through home visits or phone (if woman has one) during the next 1-2 days to screen for on-going pregnancies and assess acceptability the self-assessment.
  Other Names: Duo test
  Arms: Duo test
Other: Routine assessment — Follow up in the clinic
  Arms: Routine follow up

SUMMARY:
It is estimated that around 50 000 women die every year due to consequences of unsafe abortion (Singh et al, 2009). A majority of these deaths occur in low-income countries where access to safe abortion care is limited. Unplanned pregnancy and unsafe abortion thus place a huge burden on scarce medical resources. Any improvement in Comprehensive Abortion Care (CAC) would mean important improvements for the concerned women and their families (Singh, 2006) as well as for the societies at large. Recommended improvements concern increased access to the safest and most cost-effective methods such as medical abortion provided at primary level facilities (Singh et al, 2009). A Cochrane Review concludes that most randomised controlled trials within the field of medical abortion are conducted in high-income settings with good access to emergency health care services (Kulier et al, 2004). A simplified regime for medical abortion, which could be used at primary level facilities, would contribute to the reduction of maternal mortality and morbidity related to unsafe abortions globally. However, there is a knowledge gap in order to determine if a simplified follow up of medical abortion is equally effective as the standard procedure in a low-income setting. The results will provide evidence-based information to be used in revising training and service delivery guidelines' in order to reduce maternal mortality and morbidity in both low and high-income setting.

ELIGIBILITY:
Inclusion Criteria:

* women presenting with a positive urine test and uterine size equivalent to or up to 9 +0 weeks (63 days) of gestation
* opting for medical abortion and
* residing in an area where follow-up is feasible.
* woman agrees for a follow up contact at 10-14 days.

Exclusion Criteria:

* women with contraindications to medical abortions,
* haemoglobin level less than 85 (Hb < 85) and
* age less than 18 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Efficacy | At 10-14 days follow up
  efficacy of self-assessment, measured as the rate of complete abortion, relative to routine follow up . The percentage of women requiring surgical intervention, extra visits and administration of additional misoprostol will be used to monitor incomplete abortion.

SECONDARY OUTCOMES:
Safety | Up to 10-14 days Follow Up
  unscheduled visits for various adverse events/complications, side effects of medical abortion including infections, bleeding, pain

OTHER OUTCOMES:
contraceptive uptake | at approx. 2 weeks after abortion (at FU)
  Number of women who have started a contraceptive method or is planning to start a method
time consumption | at 10-14 days Follow Up
  Time spent for clinical visits/contacts
Acceptability | at 10-14 days follow up
  Acceptability (evaluated by a questionnaire)of home self assessment of complete pregnancy using a low sensitivity u-hCG test

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell Danielsson, MD, PhD, Principal Investigator — Karolinska Institutet; Sharad Iyengar, MD, Principal Investigator — Arth
Locations (1):
- ARTH, Udaipur, Rajasthan, India

REFERENCES:
- [Derived] Paul M, Iyengar SD, Essen B, Gemzell-Danielsson K, Iyengar K, Bring J, Klingberg-Allvin M. Does mode of follow-up influence contraceptive use after medical abortion in a low-resource setting? Secondary outcome analysis of a non-inferiority randomized controlled trial. BMC Public Health. 2016 Oct 17;16(1):1087. doi: 10.1186/s12889-016-3726-1. PMID 27745552
- [Derived] Paul M, Iyengar K, Essen B, Gemzell-Danielsson K, Iyengar SD, Bring J, Soni S, Klingberg-Allvin M. Acceptability of Home-Assessment Post Medical Abortion and Medical Abortion in a Low-Resource Setting in Rajasthan, India. Secondary Outcome Analysis of a Non-Inferiority Randomized Controlled Trial. PLoS One. 2015 Sep 1;10(9):e0133354. doi: 10.1371/journal.pone.0133354. eCollection 2015. PMID 26327217
- [Derived] Iyengar K, Paul M, Iyengar SD, Klingberg-Allvin M, Essen B, Bring J, Soni S, Gemzell-Danielsson K. Self-assessment of the outcome of early medical abortion versus clinic follow-up in India: a randomised, controlled, non-inferiority trial. Lancet Glob Health. 2015 Sep;3(9):e537-45. doi: 10.1016/S2214-109X(15)00150-3. PMID 26275330
- [Derived] Paul M, Iyengar K, Iyengar S, Gemzell-Danielsson K, Essen B, Klingberg-Allvin M. Simplified follow-up after medical abortion using a low-sensitivity urinary pregnancy test and a pictorial instruction sheet in Rajasthan, India--study protocol and intervention adaptation of a randomised control trial. BMC Womens Health. 2014 Aug 15;14:98. doi: 10.1186/1472-6874-14-98. PMID 25127545